CLINICAL TRIAL: NCT05942495
Title: A Pilot Study on the Effectiveness of Schema Focused Group Therapy for Persistent Anxiety and Depressive Symptoms: a Single Case Experimental Design
Brief Title: SFGT for Persistent Anxiety and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GGZ Noord-Holland-Noord (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL83423.018.22
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Depressive Symptoms; Anxiety Disorders; Persistent; Anxiety Depression
Keywords: schema therapy; group therapy
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single Case experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SFGT (Experimental): Whitin subject design with one arm; SFGT groep intervention
  Interventions: Behavioral: short-term schema focused group therapy

INTERVENTIONS:
Behavioral: short-term schema focused group therapy — There are two intervention phases. The first concerns the pre-treatment phase, which consists of five online sessions and three face-to-face sessions. The second intervention phase is the short-term SFGT. The SFGT consists of 17 weekly group sessions.

SUMMARY:
Rationale: Although there are effective treatments available for anxiety and depression, there is a large group of clients that does not benefit sufficiently from first-choice treatment. For this group of clients, no suitable alternative exists yet. One of the main hypothesis about maintaining factors is that there are underlying personality features that impede recovery. Schema focused therapy (SFT) is a transdiagnostic therapy focusing on underlying personality features. It has been proven to be an effective therapy for people with personality disorders and there are initial indications that SFT is also an effective treatment for anxiety and depressive symptoms. A short-term schema focused group therapy (SFGT) has been developed within GGZ-NHN, which is expected to benefit clients with persistent anxiety and depressive symptoms, but has not yet been studied.

Objective of the study: In the present study the effectiveness of short-term SFGT (protocol of De Jager, Burger & Groot) on (1) persistent anxiety and depressive symptoms, and (2) early maladaptive schemas (EMS), experiential avoidance and the mode of the healthy adult will be investigated.

DETAILED DESCRIPTION:
Study design: A Single Case Experimental Design (SCED), using repeated measures over four different phases.

ELIGIBILITY:
Inclusion Criteria:

* Persistent anxiety or depression symptoms (at least moderate score at the subscale depression (≥7 or anxiety ≥6 on the DASS-21).

  * History of at least one previous evidence-based therapy focused on anxiety, depression or PTSD according to the Dutch national guidelines.
  * Able to comprehend Dutch at a level sufficient to complete self-report.

Exclusion Criteria:

* Clients with severe problems that need to be addressed first, including substance abuse, psychosis, anxiety disorder, PTSD or depression that not have been treated.

  * Start of (or change in) medication which is not yet stabilized at the start of this study.
  * Psychosocial problems such as homelessness, no income or high debts which would make the clients unable to participate in a group.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Anxiety and depressive symptoms, as repeatedly measured by (an idiosyncratic set of) a self-report questionnaire; the Depression Anxiety Stress Scales-21 (DASS-21). | From baseline to follow-up, total of 37-40 weeks. We will administrate 10 items, idiosyncratically chosen. Measured once every 4 days.
  The DASS-21 consists of three subscales (Depression, Anxiety, and Stress). Each item can be rated on a scale from 0 ("Did not apply to me at all") to 3 ("Applied to me very much or most of the time"). All subscales content 7 items which makes the score range 0-21 for each subscale. Higher scores indicate the experience of more severe symptoms

SECONDARY OUTCOMES:
Early maladaptive schemas as measured with the Young Schema Questionnaire Short Form (YSQ-S3). | From baseline to follow-up, total of 37-40 weeks. Complete YSQ will be filled in 5 times during study. Two early maladpative schema's, 10 items, idiosyncratically chosen will be measured once every 16 days
  YSQ-S3 is a 90-item self-report questionnaire that measures 18 EMS (Young, 2005). The items are rated by a 6-point Likert scale ranging from "completely untrue" to "describes me perfectly". An average score is calculated for each EMS, with a range of 1-6. Higher scores indicate a stronger presence of the respective schema
Experiential avoidance as measured with the Brief Experiential Avoidance Questionnaire (BEAQ). | From baseline to follow-up, total of 37-40 weeks. BEAQ will be filled in once every 16 days
  The BEAQ is a 15 items self-report questionnaire with a likert scale ranging from 1 (strongly disagree) to 6 (strongly agree). Item scores are summed up making a range of 15-90; higher scores indicate more experiential avoidance.
Schema modi as measured with the Schema Modi Inventory (SMI) | From baseline to follow-up, total of 37-40 weeks. Complete SMI will be filled in 5 times during study. Mode of the healthy parent, 10 items, will be measured once every 16 days
  The SMI is a self-report questionnaire that will be used to measure 14 schema modes. The 118 items are rated at a 6-point scale ranging from "never or hardly ever" to "always". An average score is calculated for each mode, with a range of 1-6. Higher scores indicate a stronger presence of the specific schema mode.
Personality pathology as measured by the Level of Personality Functioning-screener brief form (LPFS-BF); | 25 weeks; before start baseline and after finishing therapy
  The LPFS-BF 2.0 is a brief 12-items self-report questionnaire to assess severity of personality pathology. Items ar rated on a 4-point Likert-scale rating "from very false or often false" to "very true or often true". Total score (range 0-36) of LPFS-BF can be divided into two subscales; self-functioning and interpersonal functioning. Lower scores indicate better adaptive functioning, whereas higher scores are indication for personality pathology.
General psychopathology as measured by the (totalscore of the) Outcome Questionnaire (OQ-45) | 37-40 weeks; OQ-45 will be filled in 5 times during study
  The OQ-45 which was developed to measure three domains central to mental health: symptom distress (SD), interpersonal relations (IR) and social role (SR) functioning. The self-report questionnaire consists of 45 items to be rated on a five-point Likert scale ranging from 0 (never) to 4 (almost always). Totalscore ranges from 0-180, a high score suggests that the client is admitting to a large number of symptoms as well as difficulties in interpersonal relationships, social role, and general quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Velthorst, PhD, Principal Investigator — GGZ Noord-Holland-Noord
Locations (1):
- Stichting GGZ Noord-Holland-Noord, Heerhugowaard, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No